CLINICAL TRIAL: NCT04662151
Title: A Phase 1b, Randomized, Blinded, Dose-Determined Study Evaluating the Safety and Tolerability Profile of Intervention With AT-100 (rhSP-D) in Preterm Neonates at High Risk for the Development of Bronchopulmonary Dysplasia (BPD)
Brief Title: A Clinical Safety Study of AT-100 (rhSP-D) in Preterm Neonates at High Risk for Bronchopulmonary Dysplasia (BPD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Airway Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AT-100/001
Record Dates: First submitted 2020-12-04; First posted 2020-12-10 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Bronchopulmonary Dysplasia
Keywords: Bronchopulmonary Dysplasia; Preterm; Neonate; Mechanical ventilation; Respiratory support; recombinant human Surfactant Protein-D (rhSP-D); intratracheal; air-sham
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Premature Birth

STUDY DESIGN:
Intervention Model Description: Phase 1b portion is a randomized, dual-armed, dose escalation study to establish the safest & most tolerated AT-100 dose tested as compared to air-sham alone.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1b open-label AT-100 (Experimental): Once daily AT-100 via intratracheal administration for up to 2 doses (initial Phase 1b dose-escalation portion) or 7 doses (latter Phase 1b highest tolerated & safety dose level tested portion).
  Interventions: Biological: AT-100
- Phase 1b open-label air-sham (Sham Comparator): Once daily air-sham via intratracheal administration for up to 2 doses (initial Phase 1b dose-escalation portion) or 7 doses (latter Phase 1b highest tolerated & safety dose level tested portion).
  Interventions: Procedure: Air-sham

INTERVENTIONS:
Biological: AT-100 — reconstituted AT-100 for intratracheal administration
  Other Names: (rhSP-D)
  Arms: Phase 1b open-label AT-100
Procedure: Air-sham — room air for intratracheal administration
  Arms: Phase 1b open-label air-sham

SUMMARY:
The purpose of this study is to determine if an investigational drug, AT-100, can reduce the occurrence of Bronchopulmonary Dysplasia (BPD) in babies born premature, as compared to babies born premature who receive an air-sham alone.

ELIGIBILITY:
Inclusion Criteria

1. Preterm neonates born between Gestional Age (GA):

   1. 25 0/7 weeks to 28 6/7 weeks in the initial dose escalation cohorts.
   2. 23 0/7 weeks to 28 6/7 weeks in the latter cohort.
2. Intubated and on mechanical ventilation.
3. Receiving at least 1 dose of standard-of-care-indicated surfactant treatment (Curosurf®) after birth, and able to receive the first dose of AT-100 or air-sham within 96 hours of birth given at any time point after 15 minutes following any of the subject's Curosurf® dose(s).
4. Parent or legal guardian is able to provide informed consent.

Exclusion Criteria:

1. Weight at time of birth < 400 g or > 1,800 g.
2. Major apparent congenital abnormalities impacting cardio and pulmonary function.
3. Active DNR (Do Not Resuscitate) order in place.
4. Known pulmonary air leaks (e.g. pneumothorax and pneumomediastinum) at the time of AT-100 or air-sham administration.
5. History of allergy or sensitivity to any surfactant or any component of the Investigational Product (AT-100).
6. AT-100 or air-sham dosing was set to occur before Data Safety Monitoring Committee recommendation to proceed to the next dose-escalation cohort.
7. Use of minimally invasive surfactant techniques (e.g., LISA, MIST) or INSURE or if, in the opinion of the care team, the infant is very likely too be extubated shortly after receiving Curosurf®.

   a. Subjects extubated and re-intubated after their Curosurf® dose(s) are eligible, so long as the subject meets Inclusion #3.
8. Birth mother:

   1. Has known active Hepatitis B, C, or E diagnosis.
   2. Has a known illness or exposure that, in the judgement of the Investigator, is serious enough to induce an immune deficiency such as Human Immunodeficiency Virus (HIV) and/or is receiving chemotherapy.
   3. Has known active Sexually Transmitted Infection (STI).
   4. Has known Cytomegalovirus (CMV) active infection.
   5. Has known history or evidence of alcohol or drug abuse, wit the exception of marijuana/marijuana-based products/THC, based on a positive maternal or infant drug screen as evidenced by the institution's standard-of-care practice.
9. Concurrent enrollment in an investigational drug, device, or treatment modulation trial that utilizes treatments outside of standard-of-care.
10. Any condition or situation which, in the Investigator's judgement, puts the mother or the neonate at significant risk, could confound the trial results, or may interfere significantly with the mother's or neonate's participation in the trial.
11. Symptomatic and confirmed COVID-19 infection of the mother around the time of birth.

Ages: 0 Minutes to 96 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 37 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-08-14 (Actual); Study Completion 2024-05-29 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events | Adverse events will be followed up to Day 28 of life
  Incidence and severity of adverse events between the two treatment groups will be compared
Incidence of BPD or death | Week 36 PMA

CONTACTS AND LOCATIONS:
Overall Officials: Marc O. Salzberg, MD, Study Chair — Airway Therapeutics, Inc.
Locations (18):
- United States (9):
  - Airway Therapeutics Investigational Site, Tucson, Arizona
  - Airway Therapeutics Investigational Site, Little Rock, Arkansas
  - Airway Therapeutics Investigational Site, Los Angeles, California
  - Airway Therapeutics Investigational Site, Miami, Florida
  - Airway Therapeutics Investigational Site, Atlanta, Georgia
  - Airway Therapeutics Investigational Site, Indianapolis, Indiana
  - Airway Therapeutics Investigational Site, Boston, Massachusetts
  - Airway Therapeutics Investigational Site, Durham, North Carolina
  - Airway Therapeutics Investigational Site, Norfolk, Virginia
- Spain (9):
  - Airway Therapeutics Investigational Site, Cadiz, Andalusia
  - Airway Therapeutics Investigational Site, Barcelona, Catalonia
  - Airway Therapeutics Investigational Site, Santiago de Compostela, Galicia
  - Airway Therapeutics Investigational Site, Madrid, Madrid
  - Airway Therapeutics Investigational Site, Alicante, Valencia
  - Airway Therapeutics Investigational Site, Valencia, Valencia
  - Airway Therapeutics Investigational Site, A Coruña
  - Airway Therapeutics Investigational Site, Lleida
  - Airway Therapeutics Investigational Site, Málaga

REFERENCES:
- [Background] Thebaud B, Goss KN, Laughon M, Whitsett JA, Abman SH, Steinhorn RH, Aschner JL, Davis PG, McGrath-Morrow SA, Soll RF, Jobe AH. Bronchopulmonary dysplasia. Nat Rev Dis Primers. 2019 Nov 14;5(1):78. doi: 10.1038/s41572-019-0127-7. PMID 31727986
- [Background] Jensen EA, Dysart K, Gantz MG, McDonald S, Bamat NA, Keszler M, Kirpalani H, Laughon MM, Poindexter BB, Duncan AF, Yoder BA, Eichenwald EC, DeMauro SB. The Diagnosis of Bronchopulmonary Dysplasia in Very Preterm Infants. An Evidence-based Approach. Am J Respir Crit Care Med. 2019 Sep 15;200(6):751-759. doi: 10.1164/rccm.201812-2348OC. PMID 30995069
- [Background] Sorensen GL. Surfactant Protein D in Respiratory and Non-Respiratory Diseases. Front Med (Lausanne). 2018 Feb 8;5:18. doi: 10.3389/fmed.2018.00018. eCollection 2018. PMID 29473039
- [Background] Sato A, Whitsett JA, Scheule RK, Ikegami M. Surfactant protein-d inhibits lung inflammation caused by ventilation in premature newborn lambs. Am J Respir Crit Care Med. 2010 May 15;181(10):1098-105. doi: 10.1164/rccm.200912-1818OC. Epub 2010 Feb 4. PMID 20133924
- [Background] Ikegami M, Carter K, Bishop K, Yadav A, Masterjohn E, Brondyk W, Scheule RK, Whitsett JA. Intratracheal recombinant surfactant protein d prevents endotoxin shock in the newborn preterm lamb. Am J Respir Crit Care Med. 2006 Jun 15;173(12):1342-7. doi: 10.1164/rccm.200509-1485OC. Epub 2006 Mar 23. PMID 16556693
- [Derived] Alonso-Ojembarrena A, Poindexter B, Aleem S, Healy H, Aguar-Carrascosa M, Moliner-Calderon E, Serrano-Martin MDM, Arroyo R, Vento M. A phase 1b randomized, multicenter, dose determination trial of zelpultide alfa (recombinant human surfactant protein D) in preterm neonates at high risk of developing bronchopulmonary dysplasia. Front Pediatr. 2025 Sep 12;13:1639573. doi: 10.3389/fped.2025.1639573. eCollection 2025. PMID 41018057
- See also: Airway Therapeutics' corporate website — http://www.airwaytherapeutics.com